CLINICAL TRIAL: NCT03022669
Title: Mobile Health Strategies for Veterans With Coronary Heart Disease
Brief Title: Mobile Health Strategies for Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: John Muir Medical Center (Unknown); North Florida/South Georgia Veterans Health System (Other); North Texas Veterans Healthcare System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Park, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRI 15-455
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Coronary Heart Disease
Keywords: mobile health; veterans; cardiovascular disease; medication adherence
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text Message Group (Experimental): The "TM group" will use the VA "Annie" text messaging program to remind patients to take antiplatelet medications. The content for the text messages will be determined through preliminary focus groups that will be conducted prior to the RCT.
  Interventions: Behavioral: Text Message; Other: Website
- Application Group (Experimental): The "App group" will use a mobile application to remind patients to take antiplatelet medications. The commercially available mobile app will be selected by participants through preliminary focus groups that will be conducted prior to the RCT.
  Interventions: Behavioral: Mobile Application; Other: Website
- Website-Control (Experimental): The "Website-Control group" will will be offered the American Heart Association patient education website (My Life Check - 7 Steps To Healthy Living) and will serve as an "attention-control." The website will be offered to participants in all three groups. The "7 small steps to big changes" are to manage blood pressure, control cholesterol, reduce blood sugar, get active, eat better, lose weight, and stop smoking.
  Interventions: Other: Website

INTERVENTIONS:
Behavioral: Text Message — Annie (VA text messaging program) or mobile Health manager (private text messaging program for non-VA female participants recruited at non-VA facility)
  Arms: Text Message Group
Behavioral: Mobile Application
  Arms: Application Group
Other: Website — American Heart Association patient education website

SUMMARY:
The purpose of this study is to determine whether text messages/messaging (TM) or a mobile application (app), compared with an educational website-control provided to all Veterans, can improve adherence to antiplatelet therapy among patients following acute coronary syndrome or percutaneous coronary intervention (ACS/PCI).

DETAILED DESCRIPTION:
Adherence to antiplatelet medications is critical to prevent life threatening complications (i.e., stent thrombosis); yet rates of non-adherence range from 21-57% by 12 months. Mobile technology through TM or mobile apps is a practical and inexpensive strategy to promote behavior change and enhance medication adherence. The three specific aims of this proposal are to: 1) determine preferences for content and frequency of TM to promote medication adherence through focus groups; 2) determine the most patient-centered app to promote adherence through a content analysis of all commercially available apps for medication adherence and focus groups centered on usability; and 3) compare adherence to antiplatelet medications in 225 Veterans post ACS/PCI through a randomized controlled trial. Participants will be randomized to either TM, mobile app, or website-control group. The focus groups will be stratified by low/high mobile phone use and sex.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age,
* recent ACS or PCI within 1 week
* new antiplatelet (thienopyridine) prescription
* owns a smartphone

Exclusion Criteria:

* cognitive impairment
* lack of English proficiency/literacy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in medication adherence over 12 months | 12 months
  Medication Event Monitoring System (MEMS) which is an electronic pill bottle cap that captures medication taking patterns
Change in medication adherence over 12 months | 12 months
  Adherence to Refills and Medications Scale (ARMS)- There are two subscale scores for medication taking and medication refills. The total score is found by adding both subscales. Scores can range from 12 to 48 with 12 being completely medication adherent and 48 being completely non-adherent.
Change in medication adherence at 12 months | 12 months
  Medication recall questionnaire that will assess how many missed doses there were.
Change in medication adherence at 12 months | 12 months
  VA Corporate Data Warehouse refill data (Veteran participants)
Change in medication adherence at 12 months | 12 months
  Peoplechart Meds Incontext refill data (non-Veteran participants)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Park, PhD, Principal Investigator — San Francisco Veterans Medical Center; University of California, San Francisco
Locations (5):
- United States (5):
  - John Muir Medical Center, Concord, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA North Texas Health Care System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park LG, Collins EG, Shim JK, Whooley MA. Comparing Mobile Health Strategies to Improve Medication Adherence for Veterans With Coronary Heart Disease (Mobile4Meds): Protocol for a Mixed-Methods Study. JMIR Res Protoc. 2017 Jul 18;6(7):e134. doi: 10.2196/resprot.7327. PMID 28720557